CLINICAL TRIAL: NCT01674283
Title: Effect of Glucagon on Uterine Contractility at the Time of Embryo Transfer in in Vitro Fertilization
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Uterine contractility not possible to visualize with our ultrasound machines
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVO-12-08
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Women With Fertility Disorder
MeSH Terms: interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucagon (Experimental): The first recording is a transvaginal ultrasound in midsagittale position for the measurement of the basic uterine contractility 2 minutes before the injection of Glucagon.
  The second recording is doing the same way 10 minutes after the Glucagon injection, just before the embryo transfer.
  Interventions: Drug: Glucagon
- Sodium chloride 0.9% (Placebo Comparator): The first recording is a transvaginal ultrasound in midsagittale position for the measurement of the basic uterine contractility 2 minutes before the injection of the placebo.
  The second recording is doing the same way 10 minutes after the placebo injection, just before the embryo transfer.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Glucagon
  Arms: Glucagon
Drug: placebo
  Arms: Sodium chloride 0.9%

SUMMARY:
The success of in vitro fertilization is based mainly on uterine implantation embryo. An excessive uterine contractility may interfere with implantation by a movement of the embryo in the uterus. The inhibition of the uterine contractility may have a positive effect on success rate of in vitro fertilization. It is through parenteral injection of glucagon and its spasmolytic effect on various smooth muscles and thereby on the uterine muscle, at the time of embryo transfer, the investigators intend to improve the pregnancy rates obtained after IVF.

DETAILED DESCRIPTION:
Women will have a cycle of in vitro fertilization (IVF) and follow the standard protocol established by the clinic ovo or the fertility clinic of CHUM. On the day of embryo transfer, the investigators will administer 1 mg of Glucagon or placebo intramuscularly 10 minutes before the embryo transfer. The uterine contractility will be measured by ultrasound before and after injection to document the impact of Glucagon on it and we will proceed to embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women doing fertility treatment at the clinic ovo or fertility clinic of CHUM
* Less than 40 years old
* Women with stimulate in vitro fertilization cycle
* Women able to give her consent

Exclusion Criteria:

* Body mass index > 35 kg/m2
* Women with diabetes
* Women with hypertensive disorders
* Women with a blood pressure greater or equal to 140/90 mmHg at the randomization visit
* Cons-indication to taking Glucagon:

  * Hypersensitivity to product
  * Pheochromocytoma or history of pheochromocytoma
  * Insulinoma
  * Taking a beta-blocker (drug interactions)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Uterine muscle relaxation | 30 minutes
  Determine if the intramuscular administration of 1mg of Glucagon 10 minutes before the embryo transfer is associated with a uterine muscle relaxation.

SECONDARY OUTCOMES:
Embryo implantation and pregnancy rate | 7 weeks
  Determine if the intramuscular administration of 1mg of Glucagon 10 minutes before the embryo transfer is associated with higher implantation and pregnancy rates than during embryo transfer without glucagon.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Himaya, Dr, Principal Investigator — clinique ovo and CHUM
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada